CLINICAL TRIAL: NCT03123042
Title: Feasibility Study of Sentinel Navigation Surgery in Early Gastric Cancer Patients After Non-curative Endoscopic Resection
Brief Title: Feasibility Study of Sentinel Navigation Surgery After Non-curative Endoscopic Resection
Acronym: SENORITA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Bang Wool Eom, Staff surgeon, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1710162
Record Dates: First submitted 2017-04-10; First posted 2017-04-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Sentinel Lymph Node; Early Gastric Cancer
Keywords: Sentinel lymph node; Early gastric cancer; Non-curative endoscopic resection
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentinel basin dissection (Experimental): Intervention: Sentinel basin dissection
  Interventions: Procedure: Sentinel basin dissection

INTERVENTIONS:
Procedure: Sentinel basin dissection — Sentinel basin detection using endoscopic detector (Tc99m plus indocyanine green) injection and laparoscopic sentinel basin dissection. Then conventional gastrectomy

SUMMARY:
Purpose: To prove the feasibility of sentinel node navigation surgery (SNNS) in early gastric cancer patients with the risk of lymph node metastasis after endoscopic resection and preparation of multicenter phase 3 trial of stomach preserving surgery in these patients.

Contents: The number of enrollment is 247 patients. The patients underwent endoscopic resection for early gastric cancer, and the tumor was defined to be out of indication for endoscopic resection pathologically. So, additional gastrectomy is recommended for them.

The investigators will enroll patients who agree this study. After general anesthesia, Tc99m-Phytate with indocyanine green will be injected with endoscopy. Then sentinel basin will be detected using gamma probe and laparoscopic basin dissection will be done. Sentinel lymph node will be identify in back table dissection, and patients will undergo conventional gastrectomy. Detection rate and false negative rate will be evaluated by pathological review.

DETAILED DESCRIPTION:
Sentinel basin dissection method

1. endoscopic tracer injection after general anesthesia
2. Tracer : Tc99m-phytate 3cc and indocyanine green 3cc mix --> Injection of the probe (1cc/site, 4 sites) around endoscopic submucosal dissection ulcer scar
3. Sentinel basin identification with laparoscopic probe
4. Dissection of the sentinel basin
5. Sentinel node dissection at back table
6. Conventional laparoscopic gastrectomy

ELIGIBILITY:
Inclusion Criteria:

* No limitation for age if the patient is available for gastrectomy
* Patient who underwent endoscopic submucosal dissection and the tumor was defined as out of indication.

The expanded criteria for endoscopic resection are as follows

* criterion I: intramucosal tumor without ulcerative findings and of differentiated type with size > 2 cm
* criterion II: intramucosal tumor with ulcerative findings and of differentiated type with size ≤ 3 cm
* criterion III: intramucosal tumor without ulcerative findings and of undifferentiated type with size < 2 cm
* criterion IV, submucosal invasion < 500 mm and of differentiated type with size ≤ 3 cm)
* Eastern Cooperative Oncology Group (ECOG) performance scale 0 or 1

Exclusion Criteria:

* Inoperative due to severe cardiovascular or pulmonary disease
* Pregnant
* Patients who had previous gastric surgery
* Patients who had previous upper abdomen surgery except cholecystectomy, or radiation therapy on upper abdomen, or hypersensitivity to any medicine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
detection rate (%) | 15 days after operation
  number of patients whose sentinel nodes are detected / enrolled number of patients *100

SECONDARY OUTCOMES:
False negative rate | 15 days after operation
  number of patients without metastatic lymph node in sentinel basin / number of patients with metastatic lymph node *100

CONTACTS AND LOCATIONS:
Overall Officials: Bang Wool Eom, MD, PhD, Principal Investigator — National Cancer Center, Korea
Locations (9):
- South Korea (9):
  - Bang Wool Eom, Goyang-si, Gyeonggi-do
  - Soonchunhyang University College of Medicine, Bucheon-si
  - Dongnam Institute of Radiological and Medical Science, Busan
  - Gyeongsang National University Changwon Hospital, Changwon
  - Kyungpook National University Medical Center, Daegu
  - Chonnam National University Hwasun Hospital, Hwasun
  - Gyeongsang National University Hospital, Jinju
  - Samsung Medical Center, Seoul
  - Ajou University School of Medicine, Suwon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eom BW, Yoon HM, Min JS, Cho I, Park JH, Jung MR, Hur H, Kim YW, Park YK, Nam BH, Ryu KW; Sentinel Node Oriented Tailored Approach (SENORITA) Study Group. Prospective Multicenter Feasibility Study of Laparoscopic Sentinel Basin Dissection after Endoscopic Submucosal Dissection for Early Gastric Cancer: SENORITA 2 Trial Protocol. J Gastric Cancer. 2019 Jun;19(2):157-164. doi: 10.5230/jgc.2019.19.e12. Epub 2019 Apr 15. PMID 31245160